CLINICAL TRIAL: NCT02259647
Title: Sorafenib Plus Vitamin K1 Versus Sorafenib in Advanced Hepatocellular Carcinoma - a Randomized Controlled Trial
Brief Title: Sorafenib Plus Vitamin K1 Versus Sorafenib in Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-HCC-02
Record Dates: First submitted 2014-09-11; First posted 2014-10-08 (Estimated); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sorafenib +intravenous infusion ofVit K1 (Experimental): Sorafenib 400mg twice daily + intravenous infusion ofVit K1 50 mg/day with daily increase of dose by 50 mg for 6 days, followed by oral Vitamin K1 20mg twice daily for 3month
  Interventions: Drug: Sorafenib 400mg twice daily + intravenous infusion ofVit K1
- Sorafenib+Placebo (Active Comparator): Sorafenib 400 mg twice daily + Intravenousinfusion of placebo daily for 6 days, followed by oral placebo twice daily till 3month
  Interventions: Drug: Sorafenib 400 mg twice daily + Intravenousinfusion of placebo

INTERVENTIONS:
Drug: Sorafenib 400mg twice daily + intravenous infusion ofVit K1 — Sorafenib 400mg twice daily + intravenous infusion ofVit K1 50 mg/day with daily increase of dose by 50 mg for 6 days, followed by oral Vitamin K1 20mg twice daily for 3month
  Arms: Sorafenib +intravenous infusion ofVit K1
Drug: Sorafenib 400 mg twice daily + Intravenousinfusion of placebo — Sorafenib 400 mg twice daily + Intravenousinfusion ofplacebo daily for 6 days, followed by oral placebo twice daily x 3month
  Arms: Sorafenib+Placebo

SUMMARY:
60 patients of radiological, biopsy proven advanced HCC (Hepatocellular carcinoma) patient will be randomized into two groups. Cases group will receive Sorafenib plus vitamin K and control group will receive Sorafenib plus placebo

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Child A and B cirrhosis with hepatocellular carcinoma
* Biochemical, Radiological, histological evidence of advanced hepatocellular carcinoma diagnosed as stage C and stage d with serum bilirubin <5 mg/dl according to BCLC staging system
* HCC with portal vein thrombosis
* Unresectable cancer, as assessed carefully by individual experts
* No recent active treatment like surgery, radiofrequency ablation, trans arterial chemo embolization, radiotherapy, chemotherapy (within the past 6 months)

Exclusion Criteria:

* Patients with end-stage hepatocellular carcinoma (Stage D, BCLC)with poor performance status
* Child C cirrhosis with HCC (Hepatocellular carcinoma)
* HCC with acute decompensated state of CLD - GI bleed, increased jaundice, HE, SBP (Spontaneous Bacterial Peritonitis)
* Acute febrile illness
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 1 Year

SECONDARY OUTCOMES:
Objective response rate (ORR) of tumour based on mRECIST (Response Evaluation Criteria In Solid Tumors ) criteria | 3 months
  ORR (Objective response rate) as the percentage of randomly assigned patients with complete response or partial response based on mRECIST (Response Evaluation Criteria In Solid Tumors ) criteria
Disease control rate (DCR) of tumour based on mRECIST (Response Evaluation Criteria In Solid Tumors ) criteria | 3 months
  DCR (Disease control rate) as the percentage of randomly assigned patients with complete response, partial response, or stable disease based on mRECIST (Response Evaluation Criteria In Solid Tumors ) criteria.
Biochemical response - improvement in tumor biomarker level | 3 months
Safety | 1 Years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India